CLINICAL TRIAL: NCT01776580
Title: The Association of Pelvic Organ Prolapse Severity and Urinary Symptoms and Sexual Function
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201107060RC
Record Dates: First submitted 2013-01-18; First posted 2013-01-28 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Pelvic Organ Prolapse; Sexual Dysfunction; Lower Urinary Tract Symptoms
Keywords: Pelvic organ prolapse; lower urinary tract symptoms; sexual dysfunction
MeSH Terms: conditions — Pelvic Organ Prolapse; Sexual Dysfunction, Physiological; Lower Urinary Tract Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lower urinary tract symptoms: Women with lower urinary tract symptoms

SUMMARY:
Women with pelvic organ prolapse often accompany with urinary symptoms or sexual dysfunction, and analyzing the association will be helpful to identify the indication of proper management. Therefore, the aim of this study is to identify the above associations by perineal sonography.

DETAILED DESCRIPTION:
Women with pelvic organ prolapse often accompany with urinary symptoms or sexual dysfunction, and analyzing the association will be helpful to identify the indication of proper management. Therefore, the aim of this study is to identify the above associations by perineal sonography.

ELIGIBILITY:
Inclusion Criteria:

* all patients with lower urinary tract symptoms and will undergo urodynamic studies

Exclusion Criteria:

* none

Ages: 20 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with lower urinary tract symptoms
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2011-07; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
To assess the correlation of bladder descent and lower urinary tract symptoms. | 1 day
  To assess the correlation of bladder descent and lower urinary tract symptoms, and identify which symptoms is best correlated with bladder descent during Valsalva maneuver.

SECONDARY OUTCOMES:
To identify the correlation of bladder descent with sexual dysfunction. | 1 year
  To identify which parameters of sexual dysfunction is best correlated with the bladder descent.

CONTACTS AND LOCATIONS:
Overall Officials: Ho-Hsiung Lin, MD, PhD, Principal Investigator — Department of Obstetrics & Gynecology, National Taiwan University Hospital
Locations (1):
- Department of Obstetrics & Gynecology, National Taiwan University Hospital, Taipei, Taiwan, Taiwan